CLINICAL TRIAL: NCT02648451
Title: Tolerance and Acceptability of AYMES ROME
Brief Title: Acceptability and Tolerance Study of New Oral Nutritional Supplement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aymes International Limited (Industry)
Collaborators: Alison Clark Health and Nutrition (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AY:SJ1
Record Dates: First submitted 2015-12-18; First posted 2016-01-07 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- intervention (Experimental): Patients established on an oral nutritional supplement, being prescribed 1-2 oral nutritional supplement (ONS) providing at least 300 kcal/day will be changed onto an equivalent prescription of AYMES Rome for a period of 9 days
  Interventions: Dietary Supplement: AYMES ROME

INTERVENTIONS:
Dietary Supplement: AYMES ROME — AYMES Rome is a powder, designed to be mixed with 250 ml water to make up a juice style ONS. When made up AYMES Rome provides 300 kcal (1 kcal / ml) and 10.7 g protein. It is not designed to be used as a sole source of nutrition. It is a Food for Special Medical Purposes (FSMP) and must therefore be used under medical supervision.

SUMMARY:
* To evaluate tolerance and acceptability of AYMES ROME in patients requiring supplementary oral nutritional support compared with currently available alternatives.
* To obtain data to support a submission to Advisory Committee on Borderline Substances (ACBS) for AYMES ROME (to allow for prescription in the community at National Health Service (NHS) expense).

DETAILED DESCRIPTION:
To evaluate tolerance and acceptability of AYMES ROME in patients requiring supplementary oral nutritional support compared with currently available alternatives, measuring outcomes of GI effects, Compliance, product preference,convenience etc.

To obtain data to support an ACBS submissions for AYMES ROME (to allow for prescription in the community at NHS expense).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) who are able to communicate their views regarding acceptability.
* Patients established on an oral nutritional supplement, being prescribed 1-2 ONS providing approximately 300kcal/day
* Patients expected to require oral nutritional supplementation for at least 2 further weeks.
* Informed consent obtained.

Exclusion Criteria:

* Participation in any other studies involving investigational or marketed products concomitantly or within two weeks prior to entry into the study
* Patients requiring a milk free diet
* Patients with medical or dietary contraindication to any feed ingredients (see appendix 2 of protocol for full list)
* Patients with significant renal or hepatic impairment
* Patients with swallowing impairment requiring thickened fluids
* Patients with inflammatory bowel disease or previous bowel resection.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
GI side effects when using AYMES Rome | 9 days
  Recording of absence/presence of any nausea, vomiting, abdominal pain, bloating / flatulence, when using AYMES Rome as assessed by presence / absence of side effect compared to baseline period

SECONDARY OUTCOMES:
Change to bodyweight of subjects when using AYMES Rome | 9 days
  Recording of bodyweight (in kg) at start of study, start of intervention and end of intervention for comparison to investigate any trend in weight change during the intervention period compared to baseline
Compliance with prescription of AYMES Rome | 9 days
  Recording of amount of AYMES Rome consumed by subjects compared to amount prescribed. Good compliance = >80% of prescribed being consumed. Same data collected for baseline product and compared with that of AYMES Rome
Bowel habits of subjects when using AYMES Rome - frequency | 9 days
  Recording of bowel habits whilst subjects consuming AYMES Rome, as assessed by frequency of bowel movements (number of stools per day) and compared to same data recorded during baseline period
Bowel habits of subjects when using AYMES Rome - stool consistency | 9 days
  Recording of bowel habits whilst subjects consuming AYMES Rome, as assessed by consistency of stools (assessed by Bristol Stool Chart) and compared to same data recorded during baseline period

CONTACTS AND LOCATIONS:
Overall Officials: Alison Clarke, BSc (Hons), Principal Investigator — Alison Clark Health and Nutrition

IPD SHARING:
Plan to Share IPD: No